CLINICAL TRIAL: NCT00395369
Title: Effect of Intraoperative Aprotinin Administration on Post Cardiac Surgery Optic Nerve and Retinal Thickness.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: SOR439106CTIL
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2006-11-03 (Estimated); Status verified 2006-11

CONDITIONS: Cardiac Surgery
Keywords: aprotinin; cardiac surgery; neurological dysfunction; optical coherance tomography

INTERVENTIONS:
Drug: intraoperative aprotinin administration

SUMMARY:
Cognitive and neurological dysfunction after coronary artery bypass surgery (CABG) is common and multi-factorial in origin. Several previous studies have shown that intraoperative aprotinin administration may be neuroprotective.in the current prospective randomized study, the effect of intraoperative aprotinin administration on the integrity of the optic nerve and retinal nerve fiber layer will be examined. Optical coherance tomography will be used to examin the optic nerve and retinal nerve fiber layer.

DETAILED DESCRIPTION:
Cognitive and neurological dysfunction after coronary artery bypass surgery (CABG) is common and multi-factorial in origin. Causative factors include cerebral Embolization (1), cerebral ischemia reperfusion (2), cerebral hyperthermia after discontinuation of cardiopulmonary bypass (CPB) (3), and the systemic inflammatory response to CPB (4). Cognitive dysfunction is reported in 53% of patients at discharge from the hospital, 36% at six weeks and 42% at five years (5). Cognitive function at discharge from hospital is a predictor of long-term cognitive outcome (5). Adverse neurological outcome has been classified as: type I (focal neurological injury, stupor or coma) and type II (deterioration in intellectual function, memory deficit or seizures). Patients with adverse cerebral outcomes have greater in-hospital mortality, longer hospitalization and a greater rate of discharge to facilities for intermediate or long-term care (6). Adverse neurological outcome after otherwise successful surgery is devastating for the patient, their family and society.

Neurocognitive testing is the most established method to assess post cardiac surgery cognitive outcome. Despite the extensive use of neurocognitive testing procedures in the research literature, there is uncertainty regarding the precise interpretation of findings in any given study. Thus, new tools to evaluate cognitive outcome are now being investigated.

Aprotinin is a naturally occurring serine protease inhibitor that is being used with increasing frequency in cardiac surgery to reduce blood loss and the need for perioperative blood transfusion. Through inhibition of serine proteases such as plasmin, aprotinin significantly reduces fibrinolysis, thereby aiding hemostasis during surgical procedures. These proven benefits are supplemented by the anti-inflammatory properties of aprotinin, which may help curb some of the deleterious effects of cardiopulmonary bypass. Two aprotinin dosing regimens are used for prophylactic reduction of perioperative blood loss and the need for blood transfusion in patients undergoing cardiopulmonary bypass (CPB). Serum concentrations achieved with the full-dose regimen inhibit both kallikrein and plasmin activity resulting in attenuation of the systemic inflammatory response to bypass, whereas serum concentrations achieved with the half-dose regimen only inhibit plasmin activity.

In-spite of the fact that aprotinin has been administered for more than a decade to cardiac surgery patients, it's safety is still controversial. Several studies have reported an increase risk for postoperative MI, CVA and renal failure after it's usage. Thus, its usage is not a standard of care, and depends on the surgeon decision (13).

Evidence supporting the neuroprotective effects of aprotinin given during surgery was obtained in several studies.

In a post hoc analysis of 816 CABG patients from a multicenter study (7), aprotinin administration was associated with a significantly (P = 0.04) decreased incidence of stroke (3.1% vs. 0.0%). A meta-analysis (8) of placebo-controlled, randomized, double-blind studies of CABG patients receiving high-dose aprotinin or placebo has supported the hypothesis and reported stroke incidence of 4.2% vs. 0%. A number of prospective studies have shown reduction in post cardiac surgery cognitive deficits when aprotinin was administered during CPB (9-10).

Although, the mechanism by which aprotinin may confer neuroprotection is not known, an anti-inflammatory effect can be postulated. Another possible neuroprotective mechanism is improved recovery of cerebral metabolism after ischemia (11). Its main site of action may be the microcirculation, where it decreases ischemic injury by decreasing bradykinin generation (12) and provides a better microcirculatory environment during early reperfusion.

Processes inflicting Cerebrovascular ischemia and inflammatory damage may also affect the optic nerve. Thus, pathophysiological findings discovered by optic nerve imaging can reflect cerebrovascular status.

Ischemic damage to the optic nerve or ischemic optic neuropathy (ION) is a known complication of CABG. ION describes a defect of the optic nerve leading to irreversible loss of vision in most cases. Influenced by a variety of factors, pathophysiological microvascular changes are believed to provoke anterior ischemic neuropathy with sudden painless loss of vision. Since therapeutic trials have failed, there is no reliable and effective treatment of anterior ischemic optic neuropathy and prevention of possible causes is the only way to avoid this rare but severe complication of cardiac surgery. The following risk factors were determined for ION following CABG: History of glaucoma or other ophthalmological problems, prolonged cardiopulmonary bypass-time, myocardial ischemia, general edema during cardiopulmonary bypass, excessive hemodilution with low hemoglobin and hematocrit, hypo- or hypertension, systemic hypothermia, need for vasoactive medication, diabetes and anemia.

RNFL thickness as measured by optical coherence tomography OCT has been shown to correlate very well with optic nerve atrophy and visual function in optic neuritis14, 15. Using OCT measurements of optic nerve and retinal nerve fiber layer (RNFL) thickness and visual field testing as the primary outcome, we hypothesize that high-dose aprotinin administration would decrease the incidence and severity of optic nerve and retinal injury following CABG with CPB.

Materials and Methods:

Patients scheduled for primary CABG will be studied.

Exclusion criteria:

Preoperative:

1. Patients requiring concomitant noncoronary procedures.
2. Urgent operation.
3. Intra aortic balloon pump
4. Presence of allergy to aprotinin or bleeding diathesis.
5. Previous CVA.
6. Previous eye operation.
7. Glaucoma.
8. Retinopathy.

Postoperative:

1. Postoperative CVA.
2. Postoperative critical condition precluding safe performance of OCT examination.

Anesthesia, surgery and postoperative management Oral lorazepam 0.02 to 0.03 mg/kg will be administered to patients two hours before surgery. General anesthesia will be induced with fentanyl 15 to 20 µg/kg and ketamin. Muscle relaxation will be achieved using pancuronium 0.1 mg/kg. Before cannulation of the heart, heparin (at least 300 U/kg iv) will be administered to each patient. Additional heparin will be administered to achieve and maintain a cephalin kaolin time > 480 sec. CPB will be instituted using a hollow fibre oxygenator (--) and a 40-µm screen arterial filter ( ) with crystalloid priming and a non-pulsatile flow at 32.0 to 34.0°C. Pump prime will be consisted of lactated Ringer's solution 2000 mL, sodium bicarbonate 8.4% 50 mL and mannitol 20% 3 mL/kg. The pump flow rate will be maintained at 2.4 L/min x m-2 during aortic cross clamping. During CPB, pump flows will be adjusted to maintain mean arterial pressure at 65 to 80 mmHg and hematocrit will be maintained at 20 to 25%. Intermittent use of cardiotomy suction () (0.5-1 L flows) from pericardiotomy to closure of pericardium will be used. A cell saver device will not be used.

Myocardial protection will be by intermittent antegrade and retrograde blood cardioplegia administered via the aortic root and the coronary sinus respectively. A single aortic cross-clamp will be used to complete distal and proximal anastamosis. Aortic venting will be used in all patients. At the end of surgery, patients will be transferred to the intensive care unit, where mechanical ventilation will be continued until local criteria for weaning and tracheal extubation will be met.

Administration of study drug:

Patients will be randomized to a treatment group or placebo. In the treatment group, aprotinin will be administered, consisting of 2 x 106 KIU as a loading dose after induction of anesthesia, 2 x 106 KIU added to the CPB circuit prime, and a continuous infusion of 5 x 105 KIU•hr-1 during surgery. The infusion will be discontinued at the end of surgery. Patients and the ophthalmologist will be unaware of the study group to which each patient belong.

OCT and Visual Field measurements:

OCT measurements and visual fields examination will be performed in all patients prior to, 7 days and one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients admited for coronary artery bypass surgery

Exclusion Criteria:

Preoperative:

* Patients requiring concomitant noncoronary procedures.
* Urgent operation.
* Intra aortic balloon pump
* Presence of allergy to aprotinin or bleeding diathesis.
* Previous CVA.
* Previous eye operation.
* Glaucoma.
* Retinopathy.

Postoperative:

* Postoperative CVA.
* Postoperative critical condition precluding safe performance of OCT examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2007-12

PRIMARY OUTCOMES:
optical coherance tomography findings

CONTACTS AND LOCATIONS:
Overall Officials: Dan Abramov, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka Medical Center, Beersheba, Israel